CLINICAL TRIAL: NCT03473613
Title: Comparison of Cabergoline Versus Calcium Infusion in Ovarian Hyperstimulation Syndrome Prevention:Randomized Controlled Trial
Brief Title: Cabergoline Versus Calcium Infusion in Ovarian Hyperstimulation Syndrome Prevention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, ashraf nassif mahmoud elmantwe,MD, Assistant professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ashraf Elmantwe 1
Record Dates: First submitted 2018-02-22; First posted 2018-03-22 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Ovarian Hyperstimulation
Keywords: Calcium infusion; Cabergoline
MeSH Terms: interventions — Cabergoline; Calcium Gluconate; Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium infusion (Active Comparator): 10ml 10%calcium gluconate in 200ml normal saline solution given intravenously over thirty minutes, on ovum pick up day and continued for 4days
  Interventions: Drug: Calcium Gluconate
- Oral Cabergoline (Active Comparator): Receiving oral Cabergoline (cabergamon 0.5 milligram tablet ) from ovum pick up day and continued for 7days,once daily
  Interventions: Drug: Oral Cabergoline

INTERVENTIONS:
Drug: Oral Cabergoline — Giving oral Cabergoline tablet 0.5 milligram daily starting on ovum pick up day and continued for seven days
  Other Names: Cabergamon
  Arms: Oral Cabergoline
Drug: Calcium Gluconate — Giving 10 ml of 10 % calcium gluconate on 200 ml normal saline solution o.9% intravenously over thirty minutes starting on ovum pick up day and continued for four days
  Other Names: Calcium
  Arms: Calcium infusion

SUMMARY:
Giving oral Cabergoline or calcium infusion in women at high risk for developing ovarian hyperstimulation syndrome in context of assisted reproductive technologies aiming in its prevention

DETAILED DESCRIPTION:
Women undergoing in vitro fertilization or intracytoplasmic sperm injection whom were at high risk for developing ovarian hyperstimuation syndrome were received either oral Cabergoline.5mg tablets for 7days starting on ovum pick up day and continued for 7days or received 10ml of 10%calcium gluconate in 200ml normal saline on ovum pick up day and continued for 4days

ELIGIBILITY:
Inclusion Criteria:

* women undergoing assisted reproductive technologies whom at high risk for developing ovarian hyperstimulation syndrome as with high basal antimullerian hormone ,excess antral follicular count ,high seum estradiol on day of humian choronic gonadotrophin

Exclusion Criteria:women with other endocrinopathy as congenital adrenal hyperplasia , hyperprolactinemia,diabetes

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing assisted reproductive technologies
Enrollment: 230 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of ovarian hyperstimuation syndrome | 20 days from ovum pick up day
  Clinical condition occurred in context of assisted reproductive technologies in which there serous sacs fluid accumulation and hemoconcentration

SECONDARY OUTCOMES:
Types of ovarian hyperstimuation syndrome and severity | 20 days from ovum pick up day
  Clinical severity either mild ,moderate or severe and its type either early or late onst
Chemical pregnancy | 14 day from embryos transfer day
  Positive human chorionic Gonadotropin in blood
Clinical pregnancy | 5 week from embryos transfer day
  Intrauterine gestational sac

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf N Elmantwe, MD, Principal Investigator — Benha University
Locations (1):
- Ashraf nassif Elmantwe, Cairo, Elqalopia, Egypt

IPD SHARING:
Plan to Share IPD: No
Contact investigators